CLINICAL TRIAL: NCT06901258
Title: Genius PillBox: Pilot and Feasibility Study
Brief Title: Genius PillBox Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Rachel O'Conor, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00223484
Record Dates: First submitted 2025-03-17; First posted 2025-03-28 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-03

CONDITIONS: Older Adults (65 Years and Older)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Genius Pillbox (Experimental): Participants receive Genius Pillbox to use for 1 month
  Interventions: Behavioral: Genius Pillbox

INTERVENTIONS:
Behavioral: Genius Pillbox — Participants will be mailed a Genius Pillbox to their home address. Along with the pillbox, they will also receive a detailed written description to orient them to the Genius Pillbox. Participants will be expected to use the Genius pill box organizer daily for four weeks as part of their usual medication routine. Participants are also expected to fill the designated compartments with their daily pills.

SUMMARY:
The purpose of this study is to pilot test the how acceptable older adults find a commercially available pillbox organizer with embedded sensors and automated reminders to support medication adherence.

DETAILED DESCRIPTION:
The purpose of this study is to pilot test how acceptable older adults find a commercially available pillbox organizer with embedded sensors and automated reminders to support medication adherence. Individuals who agree to participate in the study will be provided with the pillbox organizer and asked to use the pillbox for 1 month. The pillbox contains 7 compartments with embedded sensors that detects if there is a pill present. Blinking lights and a flashing letter specifying the day of the week, are used to alert users to take their medicines. After taking the first dose, a 24-hour count down timer will begin. If the medication specified for that day is not taken within the target time the device will beep to alert the user. Participants will complete a structured interview at baseline and 1 month follow-up to assess demographic and health related information, medication adherence and how they found using the pillbox organizer. Additionally, if individuals have a family member who supports their medication use, they will be asked to complete an interview at the 1 month follow-up to understand how they found using the pillbox organizer.

ELIGIBILITY:
Primary Inclusion Criteria are for older adults who manage multi-drug regimens. Inclusion Criteria:

1. Age 60 or older
2. Taking 3 or more medications
3. Takes medications twice per day or less
4. Adequate cognitive capacity (defined as less than 2 errors on 6 item cognitive screener).

Additionally, a family member that assists with a participant's medicines can also be invited to participate. The family member eligibility criteria is:

1. Age 18 or older
2. Support family member taking 3 or medications, twice a day or less
3. Adequate cognitive capacity (defined as less than 2 errors on 6 item cognitive screener)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Acceptability of Pillbox | 1 Month
  Acceptability Questionnaire, scores range from 9-36, higher scores indicate greater acceptability.
Fidelity of Pillbox Use | 1 Month
  Individual items to assess use of pillbox over 30-day period. 3 items will quantify the degree and extent which the participant used the pillbox over the past 30 day.

SECONDARY OUTCOMES:
Medication Adherence | Baseline, 1 Month
  Extent of Medication Nonadherence Scale. 3-item questionnaire, scores range from 1-5 (lower scores indicate better medication adherence)
Medication Adherence | Baseline, 1 Month
  Patient Medication Adherence Questionnaire. 3-item questionnaire, scores are summed (range 0-3), and scores of 1 or greater = non-adherence

CONTACTS AND LOCATIONS:
Overall Officials: Rachel O'Conor, PhD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No